CLINICAL TRIAL: NCT01399307
Title: A Proof of Concept Study to Demonstrate the Effectiveness of Antria Cell Preparation Process (Ace Process) in Extraction of Stromal Vascular Fraction From Adipose Tissue
Brief Title: Extraction of Stromal Vascular Fraction and Stem Cells From Fat Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antria (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACEP001
Record Dates: First submitted 2011-07-16; First posted 2011-07-21 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Soft Tissue Mass Removal
Keywords: Stem; Cell; Antria; Adipose; Stromal; Vascular; Fraction; Shahram; Shah; Rahimian
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elective Liposuction (Other)
  Interventions: Procedure: Liposuction

INTERVENTIONS:
Procedure: Liposuction — Elective Liposuction

SUMMARY:
Human Adipose Tissue is considered as a new source for Stromal Stem Cells and offers a large therapeutic potential for many rare and common diseases that impacts millions of patients worldwide. The Stromal Vascular Fraction (SVF) of Adipose Tissue is relatively easy to extract with minimally invasive procedures such as elective liposuction in large quantities and therefore may be a cost effective source for cellular therapies in a wide range of medical specialties. In this study we aim to demonstrate the efficacy of Antria Cell Preparation Process© in obtaining human adipose derived Stromal Vascular Fraction (SVF) by performing histology, various cell counts, multiple surface marker tests and measurement of the residual amount of digestive enzymes as a safety measure for human clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Male or Female Age: 18 - 65 Scheduled for Liposuction Procedure Able to understand and provide written informed Consent

Exclusion Criteria:

Diagnosis of any of the following medical conditions:

Active malignancy (diagnosed within 5 years) except for adequately treated non-melanoma skin cancer or other non-invasive or in-situ neoplasm (e.g. cervical cancer) Active Infection Chronic use of NSAID's or Steroids On Radiotherapy or Chemotherapy agents Any other disease or condition that may alter the accuracy of study results (e.g. Severe Osteoporosis, Rheumatoid Arthritis and other autoimmune disorders)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
• To assess the success rate of our methodology in extraction of SVF from adipose tissue by performing cell count, cell viability tests and specific surface markers | one month

SECONDARY OUTCOMES:
To compare the effectiveness of 2 different digestive enzymes in randomly selected set of samples | one month
To measure the amount of residual digestive enzyme after the procedure | one month
To determine the time and cost of supply during the procedure | one month
To conclude logistic barriers (transport and testing of cells) | one month
Obtaining cultures to detect potential contamination by pathogenes | one month

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Rahimian, MD, Principal Investigator — Antria
Locations (2):
- United States (2):
  - Blair Plastic Surgery, Altoona, Pennsylvania
  - Indiana Regional Medical Center, Indiana, Pennsylvania